CLINICAL TRIAL: NCT04033393
Title: Decrement of the Dual-task Performance in Individuals With Young-onset Parkinson's Disease and the Training Effects
Brief Title: Dual-task Performance in Young-onset PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-05-005C
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Early Onset Parkinson Disease; Early Stage Parkinson Disease
Keywords: Executive function; Dual-task performance; Dual-task training
MeSH Terms: conditions — Parkinsonian Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game based dual-task training group (Experimental): Participants in dual-task training group will execute game based dual-task training with treadmill, 3 times per week for 8 weeks
  Interventions: Other: Game based dual-task training
- Treadmill training group (Active Comparator): Participants in treadmill training group will do treadmill training, 3 times per week for 8 weeks
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Game based dual-task training — Participants in the experimental group will receive game based dual-task training with a treadmill
  Arms: Game based dual-task training group
Other: Treadmill training — Participants in the control group will receive treadmill training
  Arms: Treadmill training group

SUMMARY:
This study aimed to investigate the effects of Game based dual-task training with treadmill on executive function and dual-task performance in individuals with early-onset PD and discuss the correlation between the change values of executive function and dual-task performance after training. Besides, investigate cortical activation after training.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as PD and Hoehn and Yahr stage between 1~3
* Age between 20 to 80
* Able to walk 10 m independently without an assistive device
* A score of greater than or equal to 24 on the mini-mental state examination (MMSE)
* In stable medical condition allowing participation in the testing protocol and intervention

Exclusion Criteria:

* Any comorbidity or disability other than PD that would preclude gait training
* Any uncontrolled health condition for which exercise was contraindicated
* Any neurological or orthopedic disease that might interfere with the study
* Server freezing of gait, FOG questionnaire > 15

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Dual-task walking performance | Change from baseline at 8 weeks
  To evaluate gait parameters while doing dual-task walking

SECONDARY OUTCOMES:
Single walking performance | Change from baseline at 8 weeks
  To evaluate gait parameters while doing single walking
Timed up and go test | Change from baseline at 8 weeks
  To evaluate functional walking ability
Parkinson's Disease Questionnaire 39 | Change from baseline at 8 weeks
  To evaluate the quality of life
Frontal lobe battery test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Trail-making test | Change from baseline at 8 weeks
  To evaluate executive function
Stroop color and word test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Verbal fluency test-Chinese version | Change from baseline at 8 weeks
  To evaluate executive function
Digit span test | Change from baseline at 8 weeks
  To evaluate executive function
Dual-task costs | Change from baseline at 8 weeks
  To compare the cost between doing dual task and single task
Functional near-infrared spectroscopy | Change from baseline at 8 weeks
  To evaluate the changes of blood perfusion in frontal lobe